CLINICAL TRIAL: NCT05245279
Title: Correlation Between the Placental Perfusion Measured in the Entire Placenta and With Sonobiopsy
Brief Title: Placental Perfusion in the Entire Placenta and With Sonobiopsy by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Andrea Suranyi, Head of placenta study group, Szeged University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 120/2015
Record Dates: First submitted 2021-12-01; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Placenta Diseases
Keywords: 3-dimensional ultrasound; ultrasound; placenta; Investigation of placenta in-vivo
MeSH Terms: conditions — Placenta Diseases

STUDY DESIGN:
Intervention Model Description: A prospective cohort study was conducted among normal pregnant women recruited at 11 to 40 gestational weeks. Placental vascularization was evaluated using the 3-DPD-indices (vascularization-index (VI); flow-index (FI); vascularization-flow-index (VFI)) with the application of the sphere-technique or scanned from the entire placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal placenta-entitle (Experimental): The 3-DPD indices was measured in the entire placenta volume.
  Interventions: Diagnostic Test: 3 dimensional ultrasound investigation; Diagnostic Test: 2 dimensional ultrasound investigation
- Normal placenta-sonobyopsy (Experimental): The 3-DPD indices was measured at cord insertion in placenta by sonobiopsy
  Interventions: Diagnostic Test: 3 dimensional ultrasound investigation; Diagnostic Test: 2 dimensional ultrasound investigation

INTERVENTIONS:
Diagnostic Test: 3 dimensional ultrasound investigation — Images that contributed to the determination of placental volume and 3-DPD indices were obtained at the time of visit. All 3-D scans ultrasound measurements were performed by a Voluson 730 Expert ultrasound machine equipped with a multifrequency probe (2-5 MHz) to acquire images. Each sample was examined using 3-D rendering mode, in which the colour and gray value information was processed and combined to supply 3-D image. For laterally located placentas, the investigator positioned the transducer on a slight lateral inclination to obtain proper images. Power Doppler window was placed over the placenta to map the vascular tree from basal to chorionic plates. The 3-D static volume box was placed over the entire placenta volume. The sweep angle was set at maximum 70°. Each image was recovered from the disk in succession for processing. During gestation, the investigator recorded one sample from each patient.
Diagnostic Test: 2 dimensional ultrasound investigation — The two-dimensional (2-D) transabdominal conventional study provided data about fetal position, biometry, body movements and fetal heart rate as well as placental localization. The factorial default setting 'Obstetrics' was applied in 2-D mode.

SUMMARY:
In this study is tested the validity of placental vascular indices obtained from placenta ultrasonographic sphere biopsy and entire placenta investigation.

DETAILED DESCRIPTION:
Although, to this date, there have been a number of human placental studies that concerned the evaluation of placental 3 dimensional power Doppler vascularization with the use of VOCAL technique, but there was no one in which placental vasculature has been compared between the sonobiopsy and whole placental volume.

ELIGIBILITY:
Exclusion criteria:

* multiple pregnancy,
* abnormal (> 3mm) nuchal translucency from 11+0 to 13+6 weeks of gestation,
* the fetal or neonatal structural or chromosomal anomaly,
* inadequate localization of the placenta (placenta praevia),
* self-reported drugs, alcohol, caffeine or nicotine abuse,
* exposed to circulatory medication (oxerutins, calcium dobesilate)
* or not signing the consent form.
* If the mother suffer from er systemic disease (e.g. diabetes, autoimmune disease, vasculitis, haemophilia, thrombophilia, HIV infection, etc)

Inclusion clriteria:

* single pregnancy
* healthy pregnant women
* no anatomical alteration of fetus
* no genetical abnormality of fetus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The investigator studed pregnat women to analise the placental funciton in-vivo.
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Maternal characteristics (BMI) | through study completion, 2 years
  The pre-pregnancy body mass index (BMI) registered at the initial visit during prenatal care was calculated as the body weight (kg) per height (m2).
Neonatal outcome 1; based on gestational age | during first day of life
  The participants were recorded by gestational age et birth
Neonatal outcome 2, based on maturation of neonates | during first day of life
  Neonates were investigatied by maturation ( gestational age before 36+6 week) (prematurity
Neonatal outcome 3, (birth weight of newborns) | during first day of life
  Neonates birth weight calculation (gram)
Neonatal outcome 4; Apgar score | during first day of life
  Neonates poor adaptation status (Apgar score (<7) at 5 minutes)
Neonatal outcome 5, (umbilical cord pH) | during first day of life
  Neonates poor adaptation status (umbilical cord pH <7.2)
Neonatal outcome 6; delivery complication | during first day of life
  Delivery complication ( cesarean section due to fetal distress)
Neonatal outcome 7, necessary of intensive care unit | during first week of life
  Neonates transfer to neonatal intensive care unit (NICU)

SECONDARY OUTCOMES:
2D ultrasound investigaiotn of gestation (fetal biometry, placentation) | during prenatal care till the labour
  Routine ultrasound examination, based on Guideline of Hungarian Obstetrics and gynecologists (fetal biometry: biparietal diameter, head circumference, abdominal circumference, femur length; investigation of the placenta, place of placentation, Grannum staging)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Wittman, Professor, Study Chair — ALBERT SZENT-GYÖRGYI CLINICAL CENTER. REGIONAL SCIENTIFIC AND RESEARCH COMMITTEE FOR HUMAN BIOLOGICAL SCIENCE.
Locations (1):
- Universitiy of Szeged, Szeged, Hungary

REFERENCES:
- [Background] Odibo AO, Zhong Y, Longtine M, Tuuli M, Odibo L, Cahill AG, Macones GA, Nelson DM. First-trimester serum analytes, biophysical tests and the association with pathological morphometry in the placenta of pregnancies with preeclampsia and fetal growth restriction. Placenta. 2011 Apr;32(4):333-8. doi: 10.1016/j.placenta.2011.01.016. Epub 2011 Feb 13. PMID 21324404
- [Background] Molnar A, Suranyi A, Jako M, Nyari T, Nemeth G. [Examination of placental three-dimensional power Doppler indices and perinatal outcome in pregnancies complicated by intrauterine growth restriction]. Orv Hetil. 2017 Jul;158(26):1008-1013. doi: 10.1556/650.2017.30784. Hungarian. PMID 28651459
- [Background] Kozinszky Z, Suranyi A, Peics H, Molnar A, Pal A. Placental Volumetry by 2-D Sonography with a New Mathematical Formula: Prospective Study on the Shell of a Spherical Sector Model. Ultrasound Med Biol. 2015 Aug;41(8):2252-8. doi: 10.1016/j.ultrasmedbio.2015.04.005. Epub 2015 May 7. PMID 25959054
- [Background] Collins SL, Stevenson GN, Noble JA, Impey L. Rapid calculation of standardized placental volume at 11 to 13 weeks and the prediction of small for gestational age babies. Ultrasound Med Biol. 2013 Feb;39(2):253-60. doi: 10.1016/j.ultrasmedbio.2012.09.003. Epub 2012 Dec 4. PMID 23219036
- [Background] Moran M, McAuliffe FM. Imaging and assessment of placental function. J Clin Ultrasound. 2011 Sep;39(7):390-8. doi: 10.1002/jcu.20846. Epub 2011 Jun 8. PMID 21656781
- [Background] Plasencia W, Akolekar R, Dagklis T, Veduta A, Nicolaides KH. Placental volume at 11-13 weeks' gestation in the prediction of birth weight percentile. Fetal Diagn Ther. 2011;30(1):23-8. doi: 10.1159/000324318. Epub 2011 Jun 23. PMID 21701132
- [Background] Merce LT, Barco MJ, Bau S. Reproducibility of the study of placental vascularization by three-dimensional power Doppler. J Perinat Med. 2004;32(3):228-33. doi: 10.1515/JPM.2004.043. PMID 15188796
- See also: Matijevic R, Kurjak A. The assessment of placental blood vessels by three-dimensional power Doppler ultrasound — https://doi.org/10.1515/JPM.2002.004
- See also: Odibo AO, Goetzinger KR, Huster KM, Christiansen JK, Odibo L, Tuuli MG. Placental volume and vascular flow assessed by 3D power Doppler and adverse pregnancy outcomes — https://doi.org/10.1016/j.placenta.2011.01.010
- See also: Tuuli MG, Houser M, Odibo L, Huster K, Macones GA, Odibo AO. Validation of placental vascular sonobiopsy for obtaining representative placental vascular indices by three-dimensional power Doppler ultrasonography — https://doi.org/10.1016/j.placenta.2009.12.018
- See also: Evaluation of placental vascularization by three-dimensional ultrasound examination in second and third trimester of pregnancies complicated by chronic hypertension, gestational hypertension or pre-eclampsia — https://doi.org/10.1016/j.preghy.2017.03.004
- See also: Demers S, Boutin A, Dembickaja R, Campanero M, Nicolaides K. Factors Associated with Placental Vascularization Measured by 3D Power Doppler Ultrasonographic Sphere Biopsy between 11 and 14 Weeks of Gestation — https://doi.org/10.1055/s-0038-1632369
- See also: Demers S, Girard M, Roberge S, Tetu A, Giguere Y, Forest J-C, et al. First-Trimester Placental and Myometrial Blood Perfusion Measured by Three-Dimensional Power Doppler in Preeclampsia — https://doi.org/10.1055/s-0034-1396686